CLINICAL TRIAL: NCT04601207
Title: A Single-center, Randomized, Double-blind, Comparator-controlled Parallel Study Investigating the Bioavailability of Cannabidiol and Δ9-Tetrahydrocannabinol in an Emulsion Product in a Healthy Population
Brief Title: A Study Investigating the Bioavailability of CBD and THC in an Emulsion Product in a Healthy Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Age Ventures LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18CBHN
Record Dates: First submitted 2020-07-29; First posted 2020-10-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Healthy; Cannabis
Keywords: Cannabis; THC; CBD; Healthy Adult
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, comparator-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solutech™- TC10 (Experimental): 10.0mg THC, 12.2 mg CBD liquid emulsion product given orally once in-clinic
  Interventions: Drug: Cannabis Preparation
- MCT-diluted Cannabis Product (Active Comparator): 10.0mg THC, 12.2 mg CBD liquid MCT-diluted oil product given orally once in-clinic
  Interventions: Drug: Cannabis Preparation

INTERVENTIONS:
Drug: Cannabis Preparation — Dosed as a single oral dose
  Other Names: Cannabis emulsion
  Arms: Solutech™- TC10
Drug: Cannabis Preparation — Dosed as a single oral dose
  Other Names: Cannabis oil
  Arms: MCT-diluted Cannabis Product

SUMMARY:
The objective of this study is to investigate the bioavailability of Cannabidiol (CBD) and Tetrahydrocannabinol (THC) in an emulsion product against a comparator product. Thirty-two participants will be randomized into a single-center, double-blind, parallel trial. Participants will be dosed in clinic and blood and urine samples will be taken over a 12-hour period. Blood and urine samples will also be collected for 48 hours post-dose at check-in visits. Questionnaires regarding drug effects and cognitive function will also be completed following each blood sampling. Participants who consumed the comparator product will be asked to return to the clinic following a wash-out period of at least 45 days to consume the emulsion product in-clinic and complete questionnaires at the same specified time points over a 12-hour period.

DETAILED DESCRIPTION:
The use of marijuana or cannabis for medicinal purposes is deeply rooted in history, and medicinal preparations from Cannabis indica and C. sativa have been used for almost 5,000 years for treating nausea, inflammation, vomiting and pain. However, the major lipophilic cannabinoids out of >60 terpenophenolic compounds that cause these effects were not identified until the early 20th century. Sativex, dronabinol, and nabilone (synthetic or similar to cannabinoids) are the only currently approved cannabis derived medicinal products in the United States and Canada for different conditions such as nausea and vomiting associated with cancer, multiple sclerosis, intractable cancer pain, etc. Controversies regarding legal, medicinal and ethical use of cannabis have increasingly placed this plant in the spotlight in recent years. Although the use of cannabis fell from favor to fear in the early 1900s, a widespread support for its use for medicinal purposes has been on the rise in several countries across the world.

Cannabidiol (CBD), a cannabinoid constituent of cannabis plants possesses anxiolytic, antipsychotic, antiemetic and anti-inflammatory properties, without exhibiting the psychoactive effects of Δ9-tetrahydrocannabinol (Δ9-THC), the other major cannabinoid from the same plant Δ9-THC and CBD are biosynthesized as Δ9-tetrahydrocannabinolic acid and cannabidiolic acid from the common precursor olivetol. Both Δ9-THC and CBD exert their effects by interacting with the G protein-coupled cannabinoid receptors (GPCRs), CB1 and CB2 with varying affinities. While CB1 receptors are expressed in large quantities in the brain and regions central nervous system, and in lower amounts in peripheral tissues; the less studied CB2 receptors have been identified to be localized to immune cells, tonsils and the spleen. The CB1 receptors have been identified to play significant roles in pain perception, memory, motor regulation, appetite, mood, and sleep, whereas the CB2 receptors have been linked with anti-inflammation, pain reduction and reducing tissue damage. Physiologically, upon activation by the endocannabinoids like anandamide and 2-arachidonylglycerol (2-AG) (which are short lived), CB1 and CB2 trigger a downstream cascade of events that mediate homeostasis and healthy functioning. In contrast, the phytocannabinoids Δ9-THC and CBD that directly or indirectly interact with CB1 and CB2 with varying affinities modulate the activities of these receptors for prolonged durations.

Δ9-THC is the major psychoactive cannabinoid and mimics the action of the endogenous cannabinoid receptor ligands anandamide and 2-AG by activating both CB1 and CB2 receptors. Due to its binding to CB1 receptors which are specifically present in the central nervous system in areas associated with pain (eg. Spinal trigeminal nucleus, amygdala, basal ganglia and periaqueductal gray), Δ9-THC possesses antinociceptive activity and is hence used as an analgesic agent in certain pain medications. In addition, Δ9-THC has also been shown to be effective in the treatment of glaucoma, nausea, chronic pain, multiple sclerosis, epilepsy and inflammation in several pre-clinical and clinical studies . However, Δ9-THC abuse is a global concern and due to the behavioural and psychological dependence, Δ9-THC has remained a subject of controversy and a largely unproved therapy with limited studies establishing its benefit-to-risk ratio, safety and efficacy for different indications.

CBD, which is the non psychoactive phytocannabinoid, and can hence be a promising therapeutic has gained increasing attention in the recent past. Previous studies have shown that CBD is a promising potential therapeutic for various disorders of the central nervous system including anxiety, epilepsy, schizophrenia, Parkinson's disease, Alzhiemer's disease, multiple sclerosis and many more. Unlike Δ9-THC, CBD does not activate CB1 and CB2, and instead blocks the cannabinoids that activate these receptors by a complex mechanism. Several groups have proposed that this activity not only results in the non-psychotropic effects exhibited by CBD but may also account for ameliorating some of the psychotropic effects shown by Δ9-THC. In addition, by lowering the psychoactivity of Δ9-THC, CBD may also potentiate some of Δ9-THC's benefits by enhancing its tolerability and widening its therapeutic window. CBD can also inhibit or delay the reuptake and hydrolysis of the endocannabinoids like anandamide and adenosine. CBD has also been hypothesized to interact with several other non-endocannabinoid signaling systems such as serotonin receptors, vanilloid receptors, GPR-55 (orphan receptors), peroxisome proliferator activated receptors (PPARs) making it a "multi-target drug". In addition to these activities, the polyphenolic ring in CBD also results in it being a potent antioxidant. All these results have prompted the exploration of the therapeutic potential of CBD for a range of neuropsychiatric as well as inflammatory disorders.

Several groups have attempted to study the pharmacokinetics and pharmacodynamics of CBD and Δ9-THC. It is generally accepted in drug research that lipophilicity promotes the passage of molecules across cellular barriers and therefore the most lipophilic compounds will have greatest intestinal absorption. Due to the lipophilicity of cannabinoids, smoking results in the fastest absorption of CBD and Δ9-THC, however, the half-life of CBD in humans was found to be between 18-33 h upon intravenous injection, 27-35 h upon smoking, and 2-5 days upon oral administration. Bioavailability of oral and smoked CBD in humans was found to be around 6% and 31%, respectively; and bioavailability of oral and smoked Δ9-THC is shown to be 4-12% and 10-27% respectively. Other studies have previously determined the time to achieve peak plasma concentration (tmax) as 1.5- 4 h for different doses of CBD and 1-2 h for different doses of Δ9-THC. This single-center, randomized, double-blind, comparator-controlled, parallel study will investigate the bioavailability of CBD and Δ9-THC in the test product- SolutechTM - TC10 manufactured by New Age Ventures LLC in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

1. Provide voluntary, written informed consent to participate in the study
2. Between 18 and 45 years of age at screening
3. Occasional users of Cannabis: Have consumed cannabis product at least once in the past 6 months and at least 4 times in their lifetime and have experienced psychotropic effects without severe adverse events (short term paranoia, belligerence, extreme hallucinations) requiring medical interventions. Eligibility will be determined on a case by case basis by the QI.
4. Must agree to a 30-day washout of cannabis products prior to baseline.
5. Willingness to complete questionnaires, records and diaries associated with the study
6. Have a Body Mass Index (BMI) in the range of 19.0 to 29.9 kg/m2 at baseline
7. Be willing to provide blood over a 12 h period via an Intravenous (IV) catheter
8. Blood pressure at screening does not exceed a systolic blood pressure (SBP) of 140 mmHg and a diastolic blood pressure (DBP) of 90 mmHg
9. Agree to refrain from smoking tobacco products, including e-cigarettes and vaporizers or consume alcohol 24 hrs prior to their baseline visit and until completion of the study period.
10. Men who are able to father children must agree to use medically acceptable methods of contraception during the study and for 30 days after the end of the study and report any pregnancies. If a subject's partner becomes pregnant during his participation in the study or within 30 days after he has completed his last drug administration, he must inform the QI immediately
11. Female participant is not of child bearing potential, which is defined as females who have had a hysterectomy or bilateral oophorectomy, bilateral tubal ligation or natural menopause (have not had menses for > 1 year, as confirmed by measurement of serum FSH ≥ 40 IU/L at screening visit) Or,

    Females of childbearing potential must agree to abstain from heterosexual intercourse or use two methods of contraception for 30 days prior to first treatment and for 30 days after the last treatment. Subjects must have a negative urine pregnancy test result at screening, baseline and visit 5. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
    * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
    * Double-barrier method
    * Intrauterine devices
    * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
    * Vasectomy of partner at least 6- months prior to screening (Female subjects whose partners who have had a vasectomy must verbally confirm that their partner's vasectomy was confirmed to be successful by previous assessment of semen samples)
12. Agree not to donate blood within 30 days after visit 2, visit 3, visit 4 and visit 5
13. Agrees to refrain from consuming supplements in section 5.3.2 during the study
14. Agrees not to drive or operate heavy machinery if feeling dizzy or drowsy following drug administration until full mental alertness is regained after treatment visits
15. Agrees to provide information of two adult contacts to be reached in the event of transportation requirements from the clinic to their home after the study visits
16. Healthy as determined by the following criteria: laboratory results, medical history, physical exam, meeting all the inclusion criteria, not meeting any of the exclusion criteria and not on any concomitant medications listed in Section 5.3. Eligibility will be assessed by the QI based on the above.

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Clinically significant abnormal laboratory results at screening as determined by the QI.
3. Verbal confirmation of hepatic or pancreatic malfunctions
4. Verbal confirmation of use of medicinal or recreational products containing CBD/THC in the past 1 month, for participants that have consumed CBD or THC containing products prior to 1 month, eligibility will be assessed by the QI on a case by case basis depending on frequency and amount.
5. Verbal confirmation of use of hemp seeds or hemp oil in the past 1 month, for participants that have consumed hemp seeds or hemp oil prior to 1 month, eligibility will be assessed by the QI on a case by case basis depending on frequency and amount.
6. Verbal confirmation of habitual use of cannabis for medical or recreational purposes: >4 times a month. For participants who have consumed cannabis products ≤4 times a month, eligibility will be assessed by the QI depending on dose and frequency of use and self reported adverse events
7. Tongue piercings and/or mouth jewelry
8. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable after an assessment by QI
9. History (within the past 5 years) of or current Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnosis of substance dependence. For participants who have a history of substance dependence greater than 5 years ago, eligibility will be assessed on a case by case basis by the QI.
10. Currently seeking or participating in treatment for substance-related disorders
11. History of participation in treatment for substance-related disorders, including successful completion of such treatment within the past 5 years. For participants who have a sought treatment for substance abuse greater than 5 years ago, eligibility will be assessed on a case by case basis by the QI.
12. Clinically significant history of or presence of any clinically significant oral or gastrointestinal pathology (e.g. mouth ulcers, chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to baseline (visit 2) and visit 5.
13. Use of prescribed or over the counter medication which in the opinion of QI will interfere with study results or safety of the subject. Please refer to Section 5.3.1 and 5.3.2.
14. Verbal confirmation of current or history of bleeding disorders. Will be assessed by QI on a case by case basis depending on the disorder
15. Participation in a clinical research trial within 30 days prior to randomization
16. Allergy or sensitivity to investigational product and MCT-diluted cannabis oil ingredients
17. Verbal confirmation of diabetes and use of diabetes medication. However, eligibility will be assessed by the QI on a case by case basis based on dose and frequency of medication.
18. Current or previous history of clinically diagnosed neuropsychiatric disorders as per qualified investigator's (QI) opinion
19. Presence of drugs: amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), nicotine (cotinine), alcohol and THC and metabolites in urine, at screening, baseline and visit 5 (if visit 5 is applicable).
20. Personal or family history (immediate family) of psychosis: including schizophrenia and affective psychosis
21. History of suicidal ideation attempts and/or behaviour
22. Individuals who are cognitively impaired and/or who are unable to give informed consent 23. Verbal confirmation of any autoimmune disease or immune-compromised (i.e. use of anti-rejection medication, rheumatoid arthritis,)

24. Positive laboratory results for HIV, Hepatitis B or C as assessed at screening.

25. Any current or recent active and unstable medical condition that could potentially affect the study objective or adversely affect the participant's ability to complete the study or safety of the subject as per the QI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC0-48h) | 48 hours (Time points assessed for AUC0-48 h: pre-dose and post-dose at 10, 20, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 and 48 hours)
  Area under the curve (AUC0-48h) for CBD, Δ9-THC, 11-OH-THC and 11-NOR-9-CARBOXY-Δ9-THC in plasma after the administration of the investigational product or active comparator product.
Maximum concentration (Cmax, 0-48h) | 48 hours (Time points assessed for AUC0-48 h: pre-dose and post-dose at 10, 20, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 and 48 hours)
  Maximum concentration (Cmax, 0-48h) for CBD, Δ9-THC, 11-OH-THC and 11-NOR-9-CARBOXY-Δ9-THC in plasma after the administration of the investigational product or active comparator product.
Time to maximum concentration (Tmax) | 48 hours (Time points assessed for AUC0-48 h: pre-dose and post-dose at 10, 20, 30, 45 minutes and 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 and 48 hours)
  Time to maximum concentration (Tmax, 0-48h) for CBD, Δ9-THC, 11-OH-THC and 11-NOR-9-CARBOXY-Δ9-THC in plasma after the administration of the investigational product or active comparator product.

SECONDARY OUTCOMES:
Urine CBD concentration | 48 hours (Time points assessed are:0 (pre-dose), 0-4, 4-8, 8-12 hours, 12-24 hours and 24-48 hours post-dose)
  CBD concentrations in urine after the acute administration of the investigational product and the active comparator product
Urine Δ9-THC concentration | 48 hours (Time points assessed are:0 (pre-dose), 0-4, 4-8, 8-12 hours, 12-24 hours and 24-48 hours post-dose)
  Δ9-THC concentrations in urine after the acute administration of the investigational product and the active comparator product
Cognitive function | 48 hours
  Assessment of cognitive functions by BrainCheck questionnaire for the investigational product and active comparator product. It involves tests of memory (immediate- and delayed-recall) and of cognitive processing and executive function (digit-symbol substitution, trail-making, Stroop Interference). Once a patient has completed the assessments, the BrainCheck platform immediately provides validated, norm-based scores to the investigators. These scores are adjusted for age, derived from a normative database ranging from ages 10 to 99. Raw scores for the different parameters are scaled and ranked in percentiles. Scores that fall within a range of one standard deviation above the mean (50th percentile) indicate "normal" cognitive function. So, overall scores above 50th percentile are graded normal cognitive function while those below 50th suggest cognitive impairment.
Subjective evaluation of drug effects | 48 hours
  This is done using the Drug-effect questionnaire (DEQ-5) which is a 5-question questionnaire evaluating the effects of the study product. The Five questions assess drug effects, perception and likability. The number and percentage of subjects per response will be presented for each time point according to treatment. Differences between groups will be assessed using a generalized linear mixed model assuming an ordinal response with treatment, time points and treatment by time points as fixed effects and subject as random effect.Outcomes will be summarized using descriptive statistics.

OTHER OUTCOMES:
Pre-emergent and post-emergent adverse events | 72 hours
  The incidence of pre-emergent and post-emergent adverse events following a single dose of the investigational product and the comparator product. Adverse events are recorded in the study diary.
Blood pressure | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on systolic and diastolic blood pressure
Heart rate | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on heart rate
Alanine aminotransferase (ALT) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on alanine aminotransferase (ALT)
Aspartate aminotransferase (AST) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on aspartate aminotransferase (AST)
Bilirubin | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on bilirubin
Creatinine | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on creatinine
Sodium ion | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on sodium ion
Potassium ion | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on potassium ion
Chloride ion | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on chloride ion
Calcium ion | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on calcium ion
Estimated glomerular filtration rate (eGFR) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on estimated glomerular filtration rate (eGFR)
White blood cell count | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on white blood cell count
Neutrophils | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on neutrophils
Lymphocytes | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on lymphocytes
Monocytes | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on monocytes
Eosinophils | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on eosinophils
Basophils | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on basophils
Red blood cell count | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on red blood cell count
Hemoglobin | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on hemoglobin
Hematocrit | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on hematocrit
Platelet count | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on platelet count
The effect of a single dose of the investigational product and the comparator product on Mean corpuscular volume (MCV) | 48 hours post dose
  Mean corpuscular volume (MCV)
Mean corpuscular hemoglobin (MCH) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on mean corpuscular hemoglobin (MCH)
Mean corpuscular hemoglobin concentration (MCHC) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on mean corpuscular hemoglobin concentration (MCHC)
Red cell distribution width (RDW) | 48 hours post dose
  The effect of a single dose of the investigational product and the comparator product on red cell distribution width (RDW)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

REFERENCES:
- [Derived] Berl V, Hurd YL, Lipshutz BH, Roggen M, Mathur EJ, Evans M. A Randomized, Triple-Blind, Comparator-Controlled Parallel Study Investigating the Pharmacokinetics of Cannabidiol and Tetrahydrocannabinol in a Novel Delivery System, Solutech, in Association with Cannabis Use History. Cannabis Cannabinoid Res. 2022 Dec;7(6):777-789. doi: 10.1089/can.2021.0176. Epub 2022 Jul 5. PMID 35787693